CLINICAL TRIAL: NCT04763226
Title: A Randomized, Double-Blinded, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986308 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Drug Effects of BMS-986308 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV021-004
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Healthy Participants
Keywords: BMS-986308; Congestive heart failure (CHF); Diuretics; Diuretic resistance; Fluid overload; Furosemide; Persistent congestion
MeSH Terms: conditions — Heart Failure; Edema | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A Furosemide (Experimental)
  Interventions: Drug: Furosemide
- Part B (SAD) (Experimental): Single Ascending Dose (SAD)
  Interventions: Drug: BMS-986308; Other: Placebo (for BMS-986308)

INTERVENTIONS:
Drug: BMS-986308 — Specified dose on specified days
  Arms: Part B (SAD)
Other: Placebo (for BMS-986308) — Specified dose on specified days
  Arms: Part B (SAD)
Drug: Furosemide — Specified dose on specified days
  Arms: Part A Furosemide

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, and drug effects of BMS-986308 compared to placebo in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must be in good health, as determined by no clinically significant deviations from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Must have a body mass index (BMI) of 18.0 kg/m^2 to 32.0 kg/m^2, inclusive, at screening. BMI = weight (kg)/height (m)^2
* Must have normal renal function at screening (and study admission) as evidenced by an estimated glomerular filtration rate (eGFR) ≥ 80 mL/min/1.73 m^2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Presence or need for urinary catheterization, urinary tract abnormality, or disorder interfering with urination
* History of tinnitus or hearing impairment, including deafness
* History or risks factors for Torsade de Pointes and Long QT syndrome (such as electrolyte imbalances, etc)
* History of, or active, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
* Consumption of caffeine or xanthine-containing food or beverages within 72 hours prior to study treatment administration
* Use of any prescription drugs or over-the-counter (OTC) acid controllers within 4 weeks prior to study treatment administration except those medications cleared by the Medical Monitor
* Use of any other drugs, including OTC medications within 1 week and herbal preparations, within 2 weeks prior to study treatment administration except those medications cleared by the Medical Monitor
* Use of diuretics (loop diuretics, thiazide diuretics, potassium-sparing diuretics [spironolactone, amiloride]), oral calcium, potassium or magnesium supplements (including multi-vitamins) or use of non-steroidal anti-inflammatory drugs within 72 hours of the first study treatment
* Use of concomitant medications that are strong inhibitors or inducers of cytochrome CYP3A4 or OATP administered within 2 weeks prior to study treatment administration and throughout the study
* Consumption of any nutrients known to modulate cytochrome P450 (CYP) enzymes activity (eg, grapefruit, or grapefruit juice,pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to first administration of study treatment
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population of healthy volunteers
* History of allergy to furosemide, sulfonamides, other loop diuretics (furosemide cohort only), BMS-986308 or related compounds, components of the suspension or solution, including hydroxypropylmethylcellulose

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 19 days
  Part B
Incidence of serious adverse events (SAEs) | Up to 19 days
  Part B
Incidence of death | Up to 19 days
  Part B
Incidence of adverse events (AEs) leading to discontinuation | Up to 19 days
  Part B
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 19 days
  Part B
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 19 days
  Part B
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 19 days
  Part B
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 19 days
  Part B
Incidence of clinically significant changes in vital signs: Supine blood pressure | Up to 19 days
  Part B
Incidence of clinically significant changes in vital signs: Heart rate | Up to 19 days
  Part B
Incidence of clinically significant changes in vital signs: Orthostatic hypotension measurements performed as per clinical research unit's standard operating procedure | Up to 19 days
  Part B
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 19 days
  Part B
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS | Up to 19 days
  Part B
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 19 days
  Part B
  The QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF | Up to 19 days
  Part B
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in cardiac telemetry | Up to 19 days
  Part B
Incidence of clinically significant changes in physical examination findings | Up to 19 days
  Part B

OTHER OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 14 days
  Part A
Incidence of serious adverse events (SAEs) | Up to 72 days
  Part A
Incidence of death | Up to 72 days
  Part A
Incidence of adverse events (AEs) leading to discontinuation | Up to 72 days
  Part A
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 14 days
  Part A
Incidence of clinically significant changes in vital signs: Supine blood pressure | Up to 14 days
  Part A
Incidence of clinically significant changes in vital signs: Heart rate | Up to 14 days
  Part A
Incidence of clinically significant changes in vital signs: Orthostatic hypotension measurements performed as per clinical research unit's standard operating procedure | Up to 3 days
  Part A
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 14 days
  Part A
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS | Up to 14 days
  Part A
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 14 days
  Part A
  The QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF | Up to 14 days
  Part A
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in cardiac telemetry | Up to 3 days
  Part A
Incidence of clinically significant changes in physical examination findings | Up to 14 days
  Part A

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm